CLINICAL TRIAL: NCT04787991
Title: A Multicenter, Open-label, ExploRatory Platform Trial to EValuate ImmunOtherapy Combinations With Chemotherapy for the Treatment of Patients With PreviousLy UnTreated MetastatIc Pancreatic AdenOcarciNoma (REVOLUTION)
Brief Title: Exploratory Platform Trial to Evaluate Immunotherapy Combinations With Chemotherapy for the Treatment of Patients With Previously Untreated Metastatic Pancreatic Adenocarcinoma
Acronym: REVOLUTION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Insight, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Cancer Research Institute, New York City (Other); Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICI0044
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Metastatic Pancreatic Adenocarcinoma; Immunotherapy; Platform study; Nivolumab; Ipilimumab; Gemcitabine; nab-paclitaxel; hydroxychloroquine; NG-350A
MeSH Terms: interventions — Nivolumab; Ipilimumab; Hydroxychloroquine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Nivolumab + Ipilimumab + nP/gem (Experimental)
  Interventions: Drug: Nivolumab (Cohort A); Drug: Ipilimumab (Cohort A, B and C); Drug: Nab-paclitaxel (nP) (Cohort A, B and C); Drug: Gemcitabine (gem) (Cohort A, B and C)
- Cohort B: Hydroxychloroquine + Ipilimumab + nP/gem (Experimental)
  Interventions: Drug: Ipilimumab (Cohort A, B and C); Drug: Hydroxychloroquine (HCQ) (Cohort B); Drug: Nab-paclitaxel (nP) (Cohort A, B and C); Drug: Gemcitabine (gem) (Cohort A, B and C)
- Cohort C: NG-350A + Ipilimumab + nP/gem (Experimental)
  Interventions: Drug: Ipilimumab (Cohort A, B and C); Drug: Nab-paclitaxel (nP) (Cohort A, B and C); Drug: Gemcitabine (gem) (Cohort A, B and C); Drug: NG350A (Cohort C)

INTERVENTIONS:
Drug: Nivolumab (Cohort A) — Nivolumab will be administered intravenously at 360 mg every 3 weeks for up to 2 years.
  Other Names: Opdivo
  Arms: Cohort A: Nivolumab + Ipilimumab + nP/gem
Drug: Ipilimumab (Cohort A, B and C) — For Cohort A and B, ipilimumab will be administered intravenously at 1mg/kg every 6 weeks for up to 2 cycles. For Cohort C, ipilimumab will be administered intravenously at 1mg/kg on C2D1 and C4D1.
  Other Names: Yervoy
Drug: Hydroxychloroquine (HCQ) (Cohort B) — Hydroxychloroquine will be administered orally daily for up to 2 years.
  Other Names: Plaquenil
  Arms: Cohort B: Hydroxychloroquine + Ipilimumab + nP/gem
Drug: Nab-paclitaxel (nP) (Cohort A, B and C) — Nab-paclitaxel will be administered intravenously at 125 mg/m2 for 2 weeks on and 1 week off, for at least 24 weeks, unless treatment discontinuation criteria are met.
  Other Names: Abraxane
Drug: Gemcitabine (gem) (Cohort A, B and C) — Gemcitabine will be administered intravenously at 1000 mg/m2 for 2 weeks on and 1 week off, for at least 24 weeks, unless treatment discontinuation criteria are met.
  Other Names: Gemzar
Drug: NG350A (Cohort C) — NG-350A will be administered intravenously on Cycle 1 Days 15 (1e12 viral particles), 17 (3e12 viral particles), and 19 (3e12 viral particles).
  Arms: Cohort C: NG-350A + Ipilimumab + nP/gem

SUMMARY:
This trial is designed to evaluate multiple clinical hypotheses and mechanistically-defined combinations to evaluate the safety and efficacy of first-line chemo-immunotherapy combinations in participants with metastatic pancreatic ductal adenocarcinoma (mPDAC).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, exploratory platform trial designed to assess the safety and antitumor activity of immunotherapy, in combination with standard of care chemotherapy, in participants with mPDAC who have not received prior therapy. Where supportive mechanistic data are available, immunotherapy may also be combined with other treatment modalities (eg, radiation). Each cohort of this platform trial will test a different immunotherapy combination and consist of up to 2 stages: an initial stage (Stage 1) to evaluate safety, biomarkers, and/or clinical activity of the combination and an expanded cohort (Stage 2), when warranted, based on the safety, clinical activity, and/or biomarker results from Stage 1. The Sponsor intends to modify and/or add new combinations to the protocol as data emerge from scientific findings, in this and other trials.

This trial will be conducted in participants with histologically or cytologically documented diagnosis of mPDAC, with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, who have not received prior systemic therapy for their disease in the metastatic setting. Participants must have adequate organ and hematologic function and acceptable performance status. Participants must consent to tumor biopsies, including a pre-treatment (baseline) and on-treatment samples.

ELIGIBILITY:
Core Inclusion Criteria

1. Participant has histologically or cytologically documented diagnosis of pancreatic adenocarcinoma with metastatic disease. Participants with locally advanced disease are not eligible.

   a. Participants with recurrent locally advanced disease are eligible, provided: i. the last dose of chemotherapy and/or radiotherapy occurred > 4 months prior to the first dose of study intervention, and; ii. no systemic or radiotherapy has been administered in the metastatic setting.
2. Participant must have measurable disease by RECIST v1.1.
3. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. A baseline tumor tissue sample is mandatory for enrollment. If archival tumor tissue is not available, then a fresh tumor biopsy must be provided.
5. Participant must be age 18 years or older.
6. Participant must have adequate organ function.

Core Exclusion Criteria

1. Participant must not have received any prior treatment, including chemotherapy, biological therapy, or targeted therapy for mPDAC, with the following exceptions and notes:

   1. Participants who have received prior neoadjuvant or adjuvant therapy for pancreatic adenocarcinoma are eligible if neoadjuvant and adjuvant therapy (including chemotherapy and/or radiotherapy) was completed more than 4 months before the start of study intervention.
   2. Prior surgical resection is permitted.
   3. Participants who have received treatment with any other enadenotucirev-based therapy or anti-CD40 antibody at any time are not eligible for the study (cohort C only).
2. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
3. Participants with an active, known or suspected autoimmune disease. Participants with: type I diabetes mellitus; hypothyroidism only requiring hormone replacement; a history of Hashimoto syndrome, within 3 years of the first dose of study intervention, which resolved to hypothyroidism alone; skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment; or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 2.5 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2.5 years
  Defined as the proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Disease control rate (DCR) | At 9 months
  Defined as the proportion of participants who achieve confirmed CR or PR or stable disease (SD) lasting at least 16 weeks
Duration of response (DOR) | Up to 2.5 years
  Defined as the time from first documentation of response (CR or PR) to first radiographic documentation of progressive disease (PD) or death due to any cause.
Progression-free survival (PFS) | Up to 2.5 years
  Defined as the time from initiation of study intervention to date of first documented radiographic progression of disease or death due to any cause.
Overall survival (OS) | Up to 2.5 years
  Defined as the time from initiation of study intervention until death due to any cause.
Overall survival (OS) at 12 months | At 12 months
  Defined as the time from initiation of study intervention until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Parker Institute for Cancer Immunotherapy, Study Director — Parker Institute for Cancer Immunotherapy
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adamska A, Domenichini A, Falasca M. Pancreatic Ductal Adenocarcinoma: Current and Evolving Therapies. Int J Mol Sci. 2017 Jun 22;18(7):1338. doi: 10.3390/ijms18071338. PMID 28640192
- [Background] Balachandran VP, Luksza M, Zhao JN, Makarov V, Moral JA, Remark R, Herbst B, Askan G, Bhanot U, Senbabaoglu Y, Wells DK, Cary CIO, Grbovic-Huezo O, Attiyeh M, Medina B, Zhang J, Loo J, Saglimbeni J, Abu-Akeel M, Zappasodi R, Riaz N, Smoragiewicz M, Kelley ZL, Basturk O; Australian Pancreatic Cancer Genome Initiative; Garvan Institute of Medical Research; Prince of Wales Hospital; Royal North Shore Hospital; University of Glasgow; St Vincent's Hospital; QIMR Berghofer Medical Research Institute; University of Melbourne, Centre for Cancer Research; University of Queensland, Institute for Molecular Bioscience; Bankstown Hospital; Liverpool Hospital; Royal Prince Alfred Hospital, Chris O'Brien Lifehouse; Westmead Hospital; Fremantle Hospital; St John of God Healthcare; Royal Adelaide Hospital; Flinders Medical Centre; Envoi Pathology; Princess Alexandria Hospital; Austin Hospital; Johns Hopkins Medical Institutes; ARC-Net Centre for Applied Research on Cancer; Gonen M, Levine AJ, Allen PJ, Fearon DT, Merad M, Gnjatic S, Iacobuzio-Donahue CA, Wolchok JD, DeMatteo RP, Chan TA, Greenbaum BD, Merghoub T, Leach SD. Identification of unique neoantigen qualities in long-term survivors of pancreatic cancer. Nature. 2017 Nov 23;551(7681):512-516. doi: 10.1038/nature24462. Epub 2017 Nov 8. PMID 29132146
- [Background] Bauer C, Kuhnemuth B, Duewell P, Ormanns S, Gress T, Schnurr M. Prevailing over T cell exhaustion: New developments in the immunotherapy of pancreatic cancer. Cancer Lett. 2016 Oct 10;381(1):259-68. doi: 10.1016/j.canlet.2016.02.057. Epub 2016 Mar 8. PMID 26968250
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Collisson EA, Bailey P, Chang DK, Biankin AV. Molecular subtypes of pancreatic cancer. Nat Rev Gastroenterol Hepatol. 2019 Apr;16(4):207-220. doi: 10.1038/s41575-019-0109-y. PMID 30718832
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Elyada E, Bolisetty M, Laise P, Flynn WF, Courtois ET, Burkhart RA, Teinor JA, Belleau P, Biffi G, Lucito MS, Sivajothi S, Armstrong TD, Engle DD, Yu KH, Hao Y, Wolfgang CL, Park Y, Preall J, Jaffee EM, Califano A, Robson P, Tuveson DA. Cross-Species Single-Cell Analysis of Pancreatic Ductal Adenocarcinoma Reveals Antigen-Presenting Cancer-Associated Fibroblasts. Cancer Discov. 2019 Aug;9(8):1102-1123. doi: 10.1158/2159-8290.CD-19-0094. Epub 2019 Jun 13. PMID 31197017
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Hellmann MD, Paz-Ares L, Bernabe Caro R, Zurawski B, Kim SW, Carcereny Costa E, Park K, Alexandru A, Lupinacci L, de la Mora Jimenez E, Sakai H, Albert I, Vergnenegre A, Peters S, Syrigos K, Barlesi F, Reck M, Borghaei H, Brahmer JR, O'Byrne KJ, Geese WJ, Bhagavatheeswaran P, Rabindran SK, Kasinathan RS, Nathan FE, Ramalingam SS. Nivolumab plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2019 Nov 21;381(21):2020-2031. doi: 10.1056/NEJMoa1910231. Epub 2019 Sep 28. PMID 31562796
- [Background] Juszczak E, Altman DG, Hopewell S, Schulz K. Reporting of Multi-Arm Parallel-Group Randomized Trials: Extension of the CONSORT 2010 Statement. JAMA. 2019 Apr 23;321(16):1610-1620. doi: 10.1001/jama.2019.3087. PMID 31012939
- [Background] Lemery S, Keegan P, Pazdur R. First FDA Approval Agnostic of Cancer Site - When a Biomarker Defines the Indication. N Engl J Med. 2017 Oct 12;377(15):1409-1412. doi: 10.1056/NEJMp1709968. No abstract available. PMID 29020592
- [Background] Looi CK, Chung FF, Leong CO, Wong SF, Rosli R, Mai CW. Therapeutic challenges and current immunomodulatory strategies in targeting the immunosuppressive pancreatic tumor microenvironment. J Exp Clin Cancer Res. 2019 Apr 15;38(1):162. doi: 10.1186/s13046-019-1153-8. PMID 30987642
- [Background] Marabelle A, Le DT, Ascierto PA, Di Giacomo AM, De Jesus-Acosta A, Delord JP, Geva R, Gottfried M, Penel N, Hansen AR, Piha-Paul SA, Doi T, Gao B, Chung HC, Lopez-Martin J, Bang YJ, Frommer RS, Shah M, Ghori R, Joe AK, Pruitt SK, Diaz LA Jr. Efficacy of Pembrolizumab in Patients With Noncolorectal High Microsatellite Instability/Mismatch Repair-Deficient Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2020 Jan 1;38(1):1-10. doi: 10.1200/JCO.19.02105. Epub 2019 Nov 4. PMID 31682550
- [Background] McAllister F, Khan MAW, Helmink B, Wargo JA. The Tumor Microbiome in Pancreatic Cancer: Bacteria and Beyond. Cancer Cell. 2019 Dec 9;36(6):577-579. doi: 10.1016/j.ccell.2019.11.004. PMID 31951558
- [Background] Morrison AH, Byrne KT, Vonderheide RH. Immunotherapy and Prevention of Pancreatic Cancer. Trends Cancer. 2018 Jun;4(6):418-428. doi: 10.1016/j.trecan.2018.04.001. Epub 2018 Apr 30. PMID 29860986
- [Background] Neoptolemos JP, Stocken DD, Friess H, Bassi C, Dunn JA, Hickey H, Beger H, Fernandez-Cruz L, Dervenis C, Lacaine F, Falconi M, Pederzoli P, Pap A, Spooner D, Kerr DJ, Buchler MW; European Study Group for Pancreatic Cancer. A randomized trial of chemoradiotherapy and chemotherapy after resection of pancreatic cancer. N Engl J Med. 2004 Mar 18;350(12):1200-10. doi: 10.1056/NEJMoa032295. PMID 15028824
- [Background] O'Hara MH, O'Reilly EM, Varadhachary G, Wolff RA, Wainberg ZA, Ko AH, Fisher G, Rahma O, Lyman JP, Cabanski CR, Mick R, Gherardini PF, Kitch LJ, Xu J, Samuel T, Karakunnel J, Fairchild J, Bucktrout S, LaVallee TM, Selinsky C, Till JE, Carpenter EL, Alanio C, Byrne KT, Chen RO, Trifan OC, Dugan U, Horak C, Hubbard-Lucey VM, Wherry EJ, Ibrahim R, Vonderheide RH. CD40 agonistic monoclonal antibody APX005M (sotigalimab) and chemotherapy, with or without nivolumab, for the treatment of metastatic pancreatic adenocarcinoma: an open-label, multicentre, phase 1b study. Lancet Oncol. 2021 Jan;22(1):118-131. doi: 10.1016/S1470-2045(20)30532-5. PMID 33387490
- [Background] Oettle H, Post S, Neuhaus P, Gellert K, Langrehr J, Ridwelski K, Schramm H, Fahlke J, Zuelke C, Burkart C, Gutberlet K, Kettner E, Schmalenberg H, Weigang-Koehler K, Bechstein WO, Niedergethmann M, Schmidt-Wolf I, Roll L, Doerken B, Riess H. Adjuvant chemotherapy with gemcitabine vs observation in patients undergoing curative-intent resection of pancreatic cancer: a randomized controlled trial. JAMA. 2007 Jan 17;297(3):267-77. doi: 10.1001/jama.297.3.267. PMID 17227978
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Riquelme E, Zhang Y, Zhang L, Montiel M, Zoltan M, Dong W, Quesada P, Sahin I, Chandra V, San Lucas A, Scheet P, Xu H, Hanash SM, Feng L, Burks JK, Do KA, Peterson CB, Nejman D, Tzeng CD, Kim MP, Sears CL, Ajami N, Petrosino J, Wood LD, Maitra A, Straussman R, Katz M, White JR, Jenq R, Wargo J, McAllister F. Tumor Microbiome Diversity and Composition Influence Pancreatic Cancer Outcomes. Cell. 2019 Aug 8;178(4):795-806.e12. doi: 10.1016/j.cell.2019.07.008. PMID 31398337
- [Background] Rosenberg A, Mahalingam D. Immunotherapy in pancreatic adenocarcinoma-overcoming barriers to response. J Gastrointest Oncol. 2018 Feb;9(1):143-159. doi: 10.21037/jgo.2018.01.13. PMID 29564181
- [Background] Rotte A. Combination of CTLA-4 and PD-1 blockers for treatment of cancer. J Exp Clin Cancer Res. 2019 Jun 13;38(1):255. doi: 10.1186/s13046-019-1259-z. PMID 31196207
- [Background] Royal RE, Levy C, Turner K, Mathur A, Hughes M, Kammula US, Sherry RM, Topalian SL, Yang JC, Lowy I, Rosenberg SA. Phase 2 trial of single agent Ipilimumab (anti-CTLA-4) for locally advanced or metastatic pancreatic adenocarcinoma. J Immunother. 2010 Oct;33(8):828-33. doi: 10.1097/CJI.0b013e3181eec14c. PMID 20842054
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Thompson FE, Midthune D, Subar AF, Kahle LL, Schatzkin A, Kipnis V. Performance of a short tool to assess dietary intakes of fruits and vegetables, percentage energy from fat and fibre. Public Health Nutr. 2004 Dec;7(8):1097-105. doi: 10.1079/PHN2004642. PMID 15548349
- [Background] Thompson FE, Midthune D, Subar AF, McNeel T, Berrigan D, Kipnis V. Dietary intake estimates in the National Health Interview Survey, 2000: methodology, results, and interpretation. J Am Diet Assoc. 2005 Mar;105(3):352-63; quiz 487. doi: 10.1016/j.jada.2004.12.032. PMID 15746822
- [Background] Vaziri-Gohar A, Zarei M, Brody JR, Winter JM. Metabolic Dependencies in Pancreatic Cancer. Front Oncol. 2018 Dec 12;8:617. doi: 10.3389/fonc.2018.00617. eCollection 2018. PMID 30631752
- [Background] Vonderheide RH. CD40 Agonist Antibodies in Cancer Immunotherapy. Annu Rev Med. 2020 Jan 27;71:47-58. doi: 10.1146/annurev-med-062518-045435. Epub 2019 Aug 14. PMID 31412220
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Yamamoto K, Venida A, Yano J, Biancur DE, Kakiuchi M, Gupta S, Sohn ASW, Mukhopadhyay S, Lin EY, Parker SJ, Banh RS, Paulo JA, Wen KW, Debnath J, Kim GE, Mancias JD, Fearon DT, Perera RM, Kimmelman AC. Autophagy promotes immune evasion of pancreatic cancer by degrading MHC-I. Nature. 2020 May;581(7806):100-105. doi: 10.1038/s41586-020-2229-5. Epub 2020 Apr 22. PMID 32376951